CLINICAL TRIAL: NCT07154602
Title: Esthetic Outcome of 3D Printed Hybrid Ceramics as Final Restorations for Single Screw Retained Implant. A Clinical Randomized Clinical Trial
Brief Title: Esthetic Outcome of 3D Printed Hybrid Ceramics as Final Restorations for Single Screw Retained Implant.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Dental Contiuing Education (Network)
Responsible Party: Principal Investigator, Ingy Ghobrial Kastour, Dr.Ingy Kastour, International Dental Contiuing Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDCE-12208025
Record Dates: First submitted 2025-08-25; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: 3D Printing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3d printed hybrid ceramic crown (Experimental): 3d printed hybrid ceramic crown for implant prosthesis in anterior and premolars maxillary teeth
  Interventions: Other: 3D printed hybrid resin ceramic crowns
- milled hybrid resin ceramic crown (Active Comparator): milled hybrid resin ceramic crown for implant prosthesis in anterior and premolar maxillary teeth
  Interventions: Other: milled hybrid resin ceramic crown

INTERVENTIONS:
Other: 3D printed hybrid resin ceramic crowns — 3D printed hybrid resin ceramic crowns in anterior and premolar maxillary teeth
  Arms: 3d printed hybrid ceramic crown
Other: milled hybrid resin ceramic crown — milled hybrid resin ceramic crown on implants in anterior and premolar maxillary teeth
  Arms: milled hybrid resin ceramic crown

SUMMARY:
clinical trial

The goal of this clinical trial is to record the esthetic outcome of the 3d printed hybrid resin crowns. It will also test which method of fabrication is advantageous than the other one. The main questions it aims to answer are:

Does any of the fabrication methods differ in its esthetic outcome?

Researcher will compare 3d printing fabrication to conventional fabrication method which is the milling technique to see if 3d printing of hybrid resin serves patients a better crown's esthetic outcome.

Participants will:

Receive a crown after implants are osseointegrated Visit the clinic once every 3 months for checkups and tests Keep records of level of patient's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 70 years old at the time of screening.
* Patients with implants placed and in need for crown restoration
* Medically free with no systemic diseases.
* Good oral hygiene with no active periodontal disease.
* Patient's having adequate interocclusal and mesiodistal restorative space for the fabrication of a single implant-supported crown.
* Patients willing and able to provide written informed consent for participation in the study, understanding its risks, benefits, and alternative treatments.

Exclusion Criteria:

* Uncontrolled systemic diseases (e.g., uncontrolled diabetes, severe cardiovascular disease, active autoimmune disorders, uncontrolled thyroid dysfunction).
* Patients with composite restoration on the labial/buccal surface implant's neighbouring.
* Immunocompromised patients or those undergoing immunosuppressive therapy.
* Patients undergoing radiation therapy to the head and neck region, or chemotherapy.
* Patients currently on or with a history of medications known to significantly affect bone metabolism (e.g., long-term bisphosphonates, corticosteroids).
* Pregnancy or lactation.
* Known allergies to titanium, resin components, or any other materials used in the study (e.g., composite, zirconia).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Aesthetic appearance | 6 months
  using visual analogue scale, patient rating from 0 to 10 where 10 is satisfied the most while 0 is least satisfied

SECONDARY OUTCOMES:
Prosthetic complications | 6 months
  Abutment fracture or crown fracture

IPD SHARING:
Plan to Share IPD: Undecided